CLINICAL TRIAL: NCT06370416
Title: A Single Arm, Exploratory Clinical Study on the Prevention of Bone Marrow Suppression Caused by Platinum Containing Chemotherapy in Advanced Non-small Cell Lung Cancer With Trilaciclib
Brief Title: the Prevention of Bone Marrow Suppression Caused by Chemotherapy in Advanced NSCLC With Trilaciclib
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yanqiu Zhao, Principal investigator, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSKY002
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer（NSCLC）; trilaciclib; Bone marrow protection; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trilaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trilaciclib group (Experimental): 240mg/m2, intravenous infusion for 30 minutes, and administration completed within 4 hours before daily chemotherapy;
  Interventions: Drug: Trilaciclib

INTERVENTIONS:
Drug: Trilaciclib — After pathological diagnosis of NSCLC, 40 eligible subjects who met the inclusion criteria were screened and given a treatment regimen of trilaciclib before chemotherapy, after signing informed consent.
  Other Names: Trilaciclib Injection

SUMMARY:
This study is a single arm, exploratory clinical study aimed at evaluating the efficacy and safety of tralazili before chemotherapy in patients with NSCLC.After pathological diagnosis of non-small cell lung cancer(NSCLC), 40 eligible subjects who met the inclusion criteria were screened and given a treatment regimen of trilaciclib before chemotherapy, after signing informed consent.

DETAILED DESCRIPTION:
This study is a single arm, exploratory clinical study aimed at evaluating the efficacy and safety of tralazili before chemotherapy in patients with non-small cell lung cancer(NSCLC).After pathological diagnosis of NSCLC, 40 eligible subjects who met the inclusion criteria were screened and given a treatment regimen of trilaciclib before chemotherapy, after signing informed consent.Record the dynamic changes in whole blood cell count; Hematological toxicity, including febrile neutropenia and associated infections; Blood product infusion and supplementation of hematopoietic raw materials; The use of hematopoietic growth factors; Systemic use of antibiotics; Score the EQ-5D-5L, FACT-L, and FACT-An scales. Perform tumor imaging evaluation according to RECIST 1.1. Baseline imaging examination should be conducted within 21 days prior to the first administration, and tumor imaging evaluation should be conducted every 6 weeks (± 7 days) since the first study drug administration, or the frequency of imaging evaluation may be increased when there are clinical indications. The imaging examination time should follow calendar days and should not be adjusted due to treatment delay or termination. Subjects who terminate the study drug treatment due to intolerable toxicity or other non disease progression reasons should continue to receive tumor evaluation follow-up until disease progression, withdrawal from the study, or death (whichever occurs earliest) Researchers will monitor potential adverse events (AEs) throughout the entire trial and grade the severity of adverse events according to the guidelines of the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) 5.0. After treatment, the subjects will undergo a 30 day safety follow-up to monitor AE. If the patient does not receive new anti-tumor treatment within 90 days after the last medication, serious adverse events (SAEs) within 90 days after the last medication will be collected. If the subject begins new anti-tumor treatment, SAEs before starting new anti-tumor treatment will be collected, whichever occurs first.

This study will be conducted in accordance with Good Clinical Practice for Drugs (GCP).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender;
* Patients with locally advanced and late stage (IIIB, IIIC, IV) NSCLC who have been confirmed by histopathology and cannot be surgically removed (without local symptoms (with or without brain metastasis)) have at least one measurable lesion that meets the RECIST 1.1 criteria
* Need to receive chemotherapy treatment (first-line chemotherapy treatment uses platinum+pemetrexed/docetaxel/albumin paclitaxel/paclitaxel; second-line chemotherapy treatment: choose the above first-line chemotherapy treatment without using chemotherapy drugs; (Note: If first-line chemotherapy treatment does not combine with immunotherapy, subsequent increase in immunotherapy patients will not be counted as an increase in the number of treatment lines, and the number of treatment lines in this trial is limited to the number of chemotherapy treatment lines)
* The laboratory inspection meets the standards
* ECOG PS score 0-1 points;
* Women: All women with potential fertility must have a negative serum pregnancy test result during the screening period, and reliable contraceptive measures must be taken 3 months after signing the informed consent form and the last dose;
* Understand and sign the informed consent form.

Exclusion Criteria:

* Diagnosed as other malignant diseases other than NSCLC within 5 years prior to initial administration (excluding curative basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curative resection of carcinoma in situ);
* Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA grade III or IV);
* Stroke or cardiovascular events within 6 months prior to enrollment
* When screening, QTcF interval>480msec, for patients with implanted ventricular pacemakers, QTcF>500msec
* Previously received hematopoietic stem cell or bone marrow transplantation
* Allergy to the investigational drug or its components;
* The researchers believe that it is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥ 3 neutropenia during chemotherapy treatment | 1-2 weeks after chemotherapy
  Neutrophils ≤ 1.0*109

SECONDARY OUTCOMES:
The incidence of grade 4 neutropenia during chemotherapy treatment | 1-2 weeks after chemotherapy
  Neutrophils ≤ 0.5*109
The incidence of grade 3 or grade 4 thrombocytopenia | 1-2 weeks after chemotherapy
  Platelets≤ 50*109
The incidence of grade 3 or 4 anemia during chemotherapy treatment | 1-3 weeks after chemotherapy
  hemoglobin<80g/L

OTHER OUTCOMES:
Objective Response Rate | every 6 weeks to 1 year
  The proportion of subjects with complete and partial remission to the total number of subjects
Disease control rate | every 6 weeks to 1 year
  The proportion of subjects with complete remission, partial remission, and stable disease among the total subjects
Progression free survival | every 6 weeks to 1 year
  The time until the first imaging disease progression or death (whichever occurs first)
Overall survival | every 90 days to 1 year
  The time from self treatment to subject's death due to any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No